CLINICAL TRIAL: NCT05889806
Title: AUD Biomarkers Study (Proteomic and Genomic Analysis of Biospecimens Involved in Diseases and Healthy Populations)
Brief Title: AUD Biomarkers Study (Proteomic and Genomic Analysis of Biospecimens)
Status: Enrolling by invitation | Type: Observational
Sponsor: Audubon Bioscience (Industry)
Responsible Party: Sponsor
Other Study IDs: US005
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Oncology; Hematologic Malignancy; Gastro-Intestinal Disorder; Autoimmune Diseases; Pregnancy Related; Infectious Disease; Cardiovascular Diseases; Genitourinary Disease; Renal Disease
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Digestive System Diseases; Autoimmune Diseases; Communicable Diseases; Cardiovascular Diseases; Urogenital Diseases; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This Study will collect leftover Specimens that are taken during standard medical care procedures (for example, tissues, whole teeth, blood, saliva, urine, fluids, and cells). Samples will first be processed for clinical purposes, and any discarded portions of the Specimen(s) will be provided to the Sponsor for the Study purposes.
  Non-Surplus Specimens Types to be Collected for Study:
  Blood Tooth Bone marrow aspirate Aqueous humor Urine Perineal specimens Rectal specimens Urethral specimens Nasal/Nasopharyngeal and throat specimens Cheek (buccal) specimens Saliva (Sputum) Oral rinse Stool samples Vaginal and cervical specimens Endometrial (uterus) samples Vaginal lavage (wash)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy subjects with no history of chronic disease
  Interventions: Other: Observational Study Only. NO Intervention.
- Subjects with various conditions: Subjects that have been diagnosed with a condition of interest such as Diabetes, NASH, Breast Cancer, Endometriosis, or other designated condition.
  Interventions: Other: Observational Study Only. NO Intervention.

INTERVENTIONS:
Other: Observational Study Only. NO Intervention. — Observational Study Only. NO Intervention.

SUMMARY:
Study purpose: to explore the entire spectrum of proteomic and genomic changes (amongst others) involved in diseases and in healthy/control populations. The Study is designed to discover biomarkers, develop and validate diagnostic assays, instruments and therapeutics as well as other medical research. Specifically, researchers may analyze proteins, RNA, DNA copy number changes, including large and small (1,000-100,000 kb) scale rearrangements, transcription profiles, epigenetic modifications, sequence variation, and sequence in both diseased tissue and case-matched germline DNA from Subjects.

DETAILED DESCRIPTION:
The primary objective of this Study is to collect high-quality tissue, whole teeth, and biofluid Specimens, and associated Clinical Data from consented Subjects.

The secondary objective of this Study is to test Specimens and associated Clinical Data to confirm pathology diagnosis and correlation of microscopic evaluation with the provided information, to assess RNA and DNA integrity or degradation, and provide overall quality control evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Subject shall be at least 18 years of age, or higher if required by Applicable Law.
2. Subject's Clinical Data shall be relevant to the Study in which he/she is participating.
3. Subject shall understand and voluntarily sign the ICF prior to the Study participation. If the Subject is illiterate, the witness must sign the ICF (see 5.6. for details). If the Subject is incapable of consenting himself/herself, the legally authorized representative must sign the ICF (see 5.6. for details).
4. Subject shall meet any other additional inclusion criteria specified in Appendices to this Protocol, or in additional written instructions of the Sponsor.
5. Subject shall be able to donate the requested Specimen(s) without compromising his/her current health status.

Exclusion Criteria:

1. Younger than 18 years of age, or higher if required by Applicable Law.
2. The individual is incapable of understanding the items listed in the ICF and the consent process unless consented by the legally authorized representative.
3. Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include willing participants that are able to provide consent (or have an LAR to provide consent on their behalf), the requested biospecimens and associated data.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2043-05-10 (Estimated); Study Completion 2043-06-10 (Estimated)

PRIMARY OUTCOMES:
Enrollment and collection totals for a diverse population of subjects/conditions involved in diseases and in healthy/control populations. | Through study completion, an average of once per year
  We will total the number of subjects and characterize the totals by disease state, gender, ethnicity and specimens contributed

CONTACTS AND LOCATIONS:
Locations (1):
- AUD, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No